CLINICAL TRIAL: NCT01969539
Title: Open Label, Non-randomised, 1-day Trial to Characterize the Performance of Two Adapter Devices Designed to Permit Use of the Respimat® Inhaler Device With Patients Requiring Mechanical Ventilation.
Brief Title: Ventilator Adapters for Combivent Respimat
Status: Terminated | Phase: Phase 4 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1012.65
Record Dates: First submitted 2013-10-14; First posted 2013-10-25 (Estimated); Results first posted 2016-02-15 (Estimated); Last update posted 2025-02-10 (Actual); Status verified 2025-01

CONDITIONS: Pulmonary Disease, Chronic Obstructive
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

ARMS (2):
- Combivent Respimat via tee adapter (Experimental): Patients (all); previously intubated and ventilated; in need of bronchodilation w/CVT-R via tee adapter
  Interventions: Drug: Combivent Respimat via tee adapter
- Combivent Respimat - ventilator adapter (Experimental): Patients (all); previously intubated and ventilated; in need of bronchodilation with /CVT-R via ventilator adapter
  Interventions: Drug: Combivent Respimat via ventilator adapter

INTERVENTIONS:
Drug: Combivent Respimat via tee adapter — Patients (all); previously intubated and ventilated; in need of bronchodilation w/CVT-R via tee adapter
  Arms: Combivent Respimat via tee adapter
Drug: Combivent Respimat via ventilator adapter — Patients (all); previously intubated and ventilated; in need of bronchodilation w/CVT-R via ventilator adapter
  Arms: Combivent Respimat - ventilator adapter

SUMMARY:
The general aim of this 1-day, open label, non-randomised, trial is to characterize the performance of two adapter devices designed to permit use of the Respimat® inhaler with patients requiring mechanical ventilation.

ELIGIBILITY:
Inclusion criteria:

* All patients or their health care proxy must sign an informed consent consistent with International Conference on Harmonization (ICH)-Good Clinical Practice (GCP) guidelines prior to participation in the trial.
* Male or female patients, 40 years of age or older
* Patients must have a pre-admission/pre-ventilation diagnosis of obstructive lung disease (emphysema, chronic bronchitis, or asthma, or a combination thereof), and have a history of treatment with an inhaled bronchodilator. Note that the availability of prior confirmatory spirometry is desirable but not required for participation in the trial
* Patients must have a clinically relevant and acceptable elective or semi-elective indication for intubation and initiation of mechanical ventilation prior to consideration for trial enrollment.

Exclusion criteria:

* Patients with disease, respiratory or non-respiratory, that is sufficiently unstable (beyond the need for intubation and routine mechanical ventilation) such that their condition will, in the opinion of the investigator (i) put them at risk because of participation in the study, (ii) influence the results of the study [including the assessment of pharmacokinetic parameters], or (iii) cause concern regarding their ability to participate in the study for its duration of one (nominal) day.
* Patients with any of the following specific conditions:

  * Any systemic or respiratory condition or degree of instability that in the judgment of the principal investigator renders the patient unlikely to safely participate in or complete the study. Investigators are encouraged to contact the trial clinical monitor or team member medicine should there be any question about the suitability of a particular patient for this study.
  * A diagnosis of thyrotoxicosis (due to the known class side effect profile of ß2-agonists)
  * A diagnosis of paroxysmal tachycardia (>100 beats per minute) (due to the known class side effect profile of ß2-agonists)
* Active/unstable cardiac ischemia

  * Unstable or life-threatening cardiac arrhythmia
  * Unstable heart failure (typically Class III or IV)
  * Renal and/or hepatic failure to an extent likely to significantly affect drug metabolism and the consequent effect on the determination of pharmacokinetic parameters as determined by the investigator.
  * Known active tuberculosis
  * Currently under treatment with chemotherapy or radiation therapy for a malignancy.
* Patients who have taken an investigational drug within one month or six half lives (whichever is greater) prior to screening. (Note that for the purpose of this trial, commercially available and previously prescribed/administered Combivent Respimat® or Combivent Metered Dose Inhaler (MDI) will not be precluded as "investigational".)
* Patients with known hypersensitivity to ß-adrenergics drugs, anticholinergic drugs, Benzalkonium chloride (BAC), Ethylenediaminetetraacetic acid (EDTA), or any other component of the Respimat® inhalation solution delivery system
* Pregnant or nursing women
* Women of childbearing potential not using two effective methods of birth control (one barrier and one non-barrier). Female patients will be considered to be of childbearing potential unless surgically sterilized by hysterectomy or bilateral tubal ligation, or post-menopausal for at least two years.However, as subjects in this study will be sedated, on mechanical ventilation for life support and under 24/7 continuous observation in the critical care setting, the use of additional birth control during the study period is not applicable.
* Patients who are currently participating in another study. Note that patients who have previously been entered into this study and have been tested with one of the two adapters are eligible for re-entry into the trial to be studied with the alternate adapter (after a minimum of 48 hours post completion of the "active" portion of the trial with the first adapter), and if all inclusion and no exclusion criteria are met.

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2013-10-14 (Actual); Primary Completion 2014-11-20 (Actual); Study Completion 2014-11-21 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Boehringer Ingelheim, Study Chair — Boehringer Ingelheim
Locations (2):
- United States (2):
  - 1012.65.00001 Boehringer Ingelheim Investigational Site, Danbury, Connecticut
  - 1012.65.00002 Boehringer Ingelheim Investigational Site, Fort Worth, Texas

IPD SHARING:
Plan to Share IPD: No
Clinical studies sponsored by Boehringer Ingelheim, phases I to IV, interventional and non-interventional, are in scope for sharing of the raw clinical study data and clinical study documents. Exceptions might apply, e.g. studies in products where Boehringer Ingelheim is not the license holder; studies regarding pharmaceutical formulations and associated analytical methods, and studies pertinent to pharmacokinetics using human biomaterials; studies conducted in a single center or targeting rare diseases (in case of low number of patients and therefore limitations with anonymization).
  For more details refer to: https://www.mystudywindow.com/msw/datatransparency

REFERENCES:
- See also: Related Info — https://www.mystudywindow.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was closed early based on the results of an interim pharmacokinetic analysis, prior to enrollment of any patient in cohort 2, therefore only the Trudell adapter was assessed (in cohort 1)
Groups:
- Combivent Respimat Via Trudell Adapter: Participants received 20 μg ipratropium bromide and 100 μg of albuterol, administered by oral inhalation via the Trudell adapter. Patients received one, two, and four puffs in a sequential order, each dose was administered 6 hours apart.
Period: Overall Study
Arm/Group | Combivent Respimat Via Trudell Adapter
Started | 11
Completed | 11
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: Treated set which included all patients who were dispensed study medication and were documented to have taken at least one dose of investigational treatment.
Arm/Group | Combivent Respimat Via Trudell Adapter
Number analyzed (Participants) | 11
Age, Continuous [Mean (Standard Deviation); unit: Years] | 70.4 (10.45)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5
  Male | 6

OUTCOME MEASURES:

1. Primary Outcome: Pre-dose Subtracted Maximum Measured Concentration of Ipratropium
Description: Pre-dose subtracted maximum measured concentration (Cmax) of ipratropium.
  Standard pharmacokinetic (PK) analyses were not conducted due to a carry-over effect. As a consequence, the pre-specified primary endpoint (maximum measured concentration of ipratropium and albuterol) was not reported. The predose subtracted Cmax was calculated instead of the primary endpoint.
Time Frame: Pre-treatment and 5 minutes (min), 15min, 30min, 60min, 2 hours (h), 4h, 6h after each inhalation of study medication
Population: Treated set
Measure: Mean (Standard Deviation); unit: pg/ml
Arm/Group | Combivent Respimat Via Trudell Adapter
Number analyzed (Participants) | 11
pg/ml
  1 puff (20/100 μg Ipr/Alb) (N=5) | 6.12 (4.1)
  2 puffs (40/200 μg Ipr/Alb) (N=9) | 12.0 (5.5)
  4 puffs (80/400 μg Ipr/Alb) (N=6) | 26.4 (11.6)

2. Secondary Outcome: Area Under the Concentration-time Curve Over the Time Interval From 0 to 6 Hour (AUC 0-6) of Ipratropium and Albuterol
Description: Area under the concentration-time curve over the time interval from 0 to 6 hour (AUC 0-6) of ipratropium and albuterol.
  This secondary endpoint was not calculated due to a carry-over effect.
Time Frame: Pre-treatment and 5 minutes (min), 15min, 30min, 60min, 2 hours (h), 4h, 6h after each inhalation of study medication
Population: Treated set
Arm/Group | Combivent Respimat Via Trudell Adapter
Number analyzed (Participants) | 0

3. Primary Outcome: Pre-dose Subtracted Maximum Measured Concentration of Albuterol
Description: Pre-dose subtracted maximum measured concentration (Cmax) of albuterol.
  Standard pharmacokinetic (PK) analyses were not conducted due to a carry-over effect. As a consequence, the pre-specified primary endpoint (maximum measured concentration of ipratropium and albuterol) was not reported. The predose subtracted Cmax was calculated instead of the primary endpoint.
Time Frame: Pre-treatment and 5 minutes (min), 15min, 30min, 60min, 2 hours (h), 4h, 6h after each inhalation of study medication
Population: Treated set
Measure: Mean (Standard Deviation); unit: ng/ml
Arm/Group | Combivent Respimat Via Trudell Adapter
Number analyzed (Participants) | 11
ng/ml
  1 puff (20/100 μg Ipr/Alb) (N=7) | 0.192 (0.352)
  2 puffs (40/200 μg Ipr/Alb) (N=10) | 0.252 (0.435)
  4 puffs (80/400 μg Ipr/Alb) (N=10) | 0.132 (0.083)

ADVERSE EVENTS:
Time Frame: From first intake of study medication until 48 hours after the last intake of study medications, 3 days
Arm/Group | Combivent Respimat Via Trudell Adapter
Serious Adverse Events (participants affected / at risk) | 0/11
Other Adverse Events (participants affected / at risk) | 0/11

LIMITATIONS AND CAVEATS:
The study was closed early based on the results of an interim pharmacokinetic analysis, prior to enrollment of any patient in cohort 2, therefore only the Trudell adapter was assessed (in cohort 1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Boehringer Ingelheim (BI) acknowledges that investigators have the right to publish the study results. Investigators shall provide BI with a copy of any publication or presentation for review prior to any submission. Such review will be done with regard to proprietary information, information related to patentable inventions, medical, scientific, and statistical accuracy within 60 days. BI may request a delay of the publication in order to protect BI's intellectual property rights.